CLINICAL TRIAL: NCT04147390
Title: Topical 0.03% Tacrolimus Versus Systemic Mycophenolate Mofetil for Preventing Graft Rejection After Repeat Keratoplasty: One-year Results of a Randomized Clinical Trial
Brief Title: Immunosuppression After Repeat Keratoplasty
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 96340
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Keratopathy
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usage mycophenolate mofetil (Active Comparator)
  Interventions: Drug: prescribe mycophenolate mofetil(MMF)
- usage tacrolimus (Active Comparator)
  Interventions: Drug: prescribe topical 0.03 % tacrolimus

INTERVENTIONS:
Drug: prescribe topical 0.03 % tacrolimus — prescribe topical 0.03 % tacrolimus 3 times a day for 12 months
  Arms: usage tacrolimus
Drug: prescribe mycophenolate mofetil(MMF) — MMF orally 1 g twice daily for the first 6 months and then 1 g daily for the next 6 months
  Arms: usage mycophenolate mofetil

SUMMARY:
Purpose: To compare the efficacy of topical 0.03% tacrolimus with systemic mycophenolate mofetil (MMF) in preventing corneal allograft rejection after repeat keratoplasty.

Design: Prospective, randomized clinical trial Introduction: Repeat keratoplasty continues to be an important indication for corneal transplantation in many centers, and it accounts for up to 41% (varying from 6% to 41%) of all keraptoplasty cases performed.

Methods: This study will enroll all patients who are candidate for repeat keratoplasty after a failed penetrating keratoplasty. Group 1 will receive MMF orally 1 g twice daily for the first 6 months and then 1 g daily for the next 6 months, and group 2 will receive topical 0.03 % tacrolimus 3 times a day for 12 months. All patients are treated with topical and oral corticosteroids postoperatively. The participants are observed closely for signs of graft rejection, and the rates of rejection-free graft survival are calculated and compared between the two groups at postoperative month 12

ELIGIBILITY:
Inclusion Criteria:

* all patients who are scheduled for repeat corneal transplantation following failed primary penetrating keratoplasty (PK )

Exclusion Criteria:

* uncontrolled increase in intraocular pressure
* active herpetic keratitis and corneal ulcer
* limbal stem cell deficiency
* a history of limbal stem cell transplantation
* age less than 18 years
* pregnancy, a history of malignant disorders
* abnormal liver or kidney function
* the presence of poorly controlled systemic hypertension
* diabetes mellitus
* systemic infections
* active peptic ulcer disease
* any gastrointestinal disorders led to patient exclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
graft rejection | 12 months
  clinical examination

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran